CLINICAL TRIAL: NCT01973361
Title: A Randomized Controlled Trial to Investigate if Application of Low Frequency Ultrasound-assisted Debridement May Improve Healing and Infection Outcomes for the Person With Vasculopathy and Recalcitrant Wounds of the Lower Extremity
Brief Title: Efficacy Study of Ultrasound-Assisted Debridement to Influence Wound Healing
Acronym: UltraHeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130152-01H
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: WOUNDS
Keywords: Wounds; Lower extremity; Diabetes; Arterial Insufficiency; Debridement; Low frequency ultrasound; Contact ultrasound; Wound clinic; Wound bed preparation; Wound infection; Chronic wound inflammation
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus; Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound debridement (Experimental): Participants receiving ultrasound assisted debridement in addition to best practice wound care.
  Interventions: Device: Ultrasound debridement
- Best Practice wound care (Active Comparator): Participants receiving best practice wound care alone
  Interventions: Device: Best practice wound care

INTERVENTIONS:
Device: Ultrasound debridement — Ultrasound-assisted wound debridement with saline irrigant applied for 5 - 15 minutes until visible and removable non-viable appearance tissue is removed to reveal a healthy appearance wound bed.
  Other Names: Misonix Sonic One Ultrasound Wound Care System
  Arms: Ultrasound debridement
Device: Best practice wound care — Participants will receive moist wound care with addition of silver alginate dressing for visual cues of infection.
  Arms: Best Practice wound care

SUMMARY:
The UltraHeal Study is a randomized controlled trial to compare healing response of low frequency contact ultrasonic-assisted debridement in addition to best practice wound care to best practice wound care alone in a Vascular Surgery Clinic patient population with wounds of the lower extremity.

DETAILED DESCRIPTION:
The study will also investigate the bacterial tissue burden and protease activity to provide further insight into the infection and inflammation aspects of healing barriers in a challenging population.

ELIGIBILITY:
Inclusion Criteria:

* Persons with lower extremity wound referred to vascular surgery service.
* Full thickness wound below the knee with surface area of at least 1cm2.
* Age >18 years
* English speaking
* Ulcer of known etiology including diabetic foot wounds, and arterial or venous leg ulcers
* Willing and able to adhere to 12 week study protocol that includes attending weekly clinic appointments, and wearing prescribed footwear or compression therapy

Exclusion Criteria:

* Leg wounds due to inflammatory conditions (e.g. pyoderma gangrenosum, vasculitis), malignancy, or other unknown etiologies.
* Severe arterial insufficiency: Absence of pedal pulses combined with Ankle Brachial Index ≤ 0.3, Toe Pressure ≤20, or Trans Cutaneous Oxygen Measure ≤20
* Presence of acute limb threatening infection
* Vascular surgery planned within next 3 months
* Exposed vascular graft or blood vessel, bone or tendon in the base of the wound.
* Currently receiving advanced wound therapy treatments: Hyperbaric therapy, biological dressings [collagen or extracellular matrix dressings].
* Increased likelihood of an adverse reaction to ultrasonic debridement due to:
* Excessive wound pain (>5 VAS scale) or patient described intolerable
* Allergy to topical anesthetic (lidocaine)
* Individuals who have factors/circumstances that are known to limit their ability to demonstrate healing in 4 weeks.

For example:

* medically unstable or palliative medical status
* poor nutritional status (low serum albumin < 15),
* anemia (Hb < 75 mg/dl),
* taking immunosuppressant medication (prednisone, chemotherapy; transplant anti-rejection medication),
* Individuals with medical conditions that contraindicate the use of ultrasound energy
* Cardiac pacemaker or defibrillator
* Excessive bleeding tendency (> 5 mins post debridement) or identified coagulopathic disorders
* Exposed bone in the wound base
* Untreated osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in wound surface area | Weekly for 4 weeks then at 12 weeks.
  The wound surface area will be measured weekly once treatment is initiated, with a final measurement 12 weeks after initiation of therapy.

SECONDARY OUTCOMES:
Protease activity | Pre-treatment, post treatment at weeks 5 and weeks then at 12 weeks.
  A wound swab to test for elevated protease activity will be obtained before treatment and at week5 (after the 4 weekly treatments), and then again at week 12 to ascertain the immediate and sustained impact on inflammatory aspects of wound healing.
Bacterial burden | Pre-treatment, week 5 and week 12
  A tissue culture to test for elevated bacterial activity and species identification will be obtained before treatment and at week 5 (after the 4 weekly treatments), and then again at week 12 to ascertain the immediate and sustained impact on infection aspects of wound healing
Number of wounds healed | Throughout duration of the study
  We will count the number of wounds that have healed and have not healed for each group and compare to ascertain if the therapy improves healing.

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Murphy, MClSc PhD(c), Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Wound Healing Centre, Ottawa, Ontario, Canada